CLINICAL TRIAL: NCT06913712
Title: Evolution of Body Mass Index in Idiopathic Intracranial Hypertension and Its Relationship With the Response to Treatment. Retrospective and Prospective Study
Brief Title: BMI in Idiopathic Intracranial Hypertension and Its Relationship With the Response to Treatment
Status: Recruiting | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Vicente Vanaclocha, Professor, University of Valencia
Other Study IDs: V 07/06/2024
Record Dates: First submitted 2025-01-12; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Intracranial Hypertension (IIH)
Keywords: Idiopathic Intracranial Hypertension; Body Mass Index; Lumboperitoneal Shunt; Ventriculoperitoneal Shunt; Acetazolamide
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Idiopathic Intracranial Hypertension: Patients with Idiopathic Intracranial Hypertension
  Interventions: Other: Weight loss without pharmacotherapy

INTERVENTIONS:
Other: Weight loss without pharmacotherapy — The study will record the weight of the patients with Idiopathic Intracranial Hypertension every three months. It will correlate with the response to the different treatment modalities (weight loss with no other intervention, diuretic drugs (acetazolamide), lumboperitoneal shunt, or ventriculoperitoneal shunt). No medication will be provided to help lose weight.

SUMMARY:
1. To establish the correlation between the evolution of the body mass index in benign intracranial hypertension and the response to treatments.
2. To establish the BMI at which this disease occurs.
3. To establish how much the BMI must be reduced to cure this disease.
4. To assess the evolution and response to treatments of sick people who DO NOT reduce or even continue to increase their BMI despite treatment with Acetazolamide or a possible CSF diversion

DETAILED DESCRIPTION:
There is unanimity that one of the causes of benign intracranial hypertension is obesity. However, there is no agreement on the upper limit of BMI above which this disease occurs or the lower limit above which it is cured. People affected by this disease often have extreme difficulty losing weight and it is not uncommon for them to have followed various diets over the years to lose weight. In general, patients prefer to take medication or to undergo surgery with the implantation of a cerebrospinal fluid diversion system that does not force them to sacrifice following a strict diet. Unfortunately, those who do not manage to lose weight noticeably present repeated complications due to malfunction of the CSF diversion system with headaches and a progressive loss of visual acuity. Among other reasons, it must be considered that cerebrospinal fluid diversion systems work by pressure gradient. Since obesity increases the pressure inside the peritoneal cavity, these shunt systems will be ineffective because they will not be able to drain even if the pressure of the shunt valve is diminished to levels below 6 mm Hg.

The aim of this study is to find out what the specific BMI goal should be for each patient in particular and to be able to make them aware of this so that they make an effort and achieve it. Patients are referred to Endocrinology to be recommended the diet to follow. In some cases, bariatric surgery is used. Still, as it does not require effort or awareness on the part of these people, it is not uncommon for them to gain weight again and for benign intracranial hypertension to recur. The usual thing is that their evolution is torpid and the repeated therapeutic attempts are fruitless or plagued by complications. Weight loss using medication such as Ozempic (Semaglutide) is not accepted internationally nor contemplated by the Endocrinology Service of the General University Hospital of Valencia. On the one hand, it has no indication and on the other hand, the possible complications are not known. In addition, patients who take it on their own initially lose weight, but when they stop taking the medication they quickly regain the lost weight as a result of not having adopted healthy eating habits.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older at the time of enrollment. There is no upper age limit to ensure inclusivity across age ranges.
* A confirmed diagnosis of Idiopathic Intracranial Hypertension, established according to the Dandy criteria.
* The diagnostic process must exclude other potential causes of increased intracranial pressure as detailed in the 'Diagnosis' section, ensuring an accurate identification of idiopathic cases.

Exclusion Criteria:

* A diagnosis other than IIH, specifically: tension-type headache, Chiari I malformation, or any other headache disorder unrelated to IIH.
* The presence of secondary causes of increased intracranial pressure (e.g., structural brain abnormalities, venous sinus thrombosis, or medication-induced factors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed to be a retrospective-prospective cohort study. Data was collected from all retrospective patients attended in the last 10 years by the Neurosurgery department at Hospital General Universitario de Valencia who presented idiopathic intracranial hypertension (IIH) and were accepted to participate. Data were extracted and reviewed from the patient's medical records.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | Through study completion, an average of 1 year
  BMI evolution in patients with benign intracranial hypertension and its relationship with the evolution of the patient's symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Consorcio Hospital General Universitario de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleinschmidt JJ, Digre KB, Hanover R. Idiopathic intracranial hypertension: relationship to depression, anxiety, and quality of life. Neurology. 2000 Jan 25;54(2):319-24. doi: 10.1212/wnl.54.2.319. PMID 10668690
- [Background] Mollan SP, Mitchell JL, Yiangou A, Ottridge RS, Alimajstorovic Z, Cartwright DM, Hickman SJ, Markey KA, Singhal R, Tahrani AA, Frew E, Brock K, Sinclair AJ. Association of Amount of Weight Lost After Bariatric Surgery With Intracranial Pressure in Women With Idiopathic Intracranial Hypertension. Neurology. 2022 Sep 13;99(11):e1090-e1099. doi: 10.1212/WNL.0000000000200839. Epub 2022 Jul 5. PMID 35790425
- [Background] Ko MW, Chang SC, Ridha MA, Ney JJ, Ali TF, Friedman DI, Mejico LJ, Volpe NJ, Galetta SL, Balcer LJ, Liu GT. Weight gain and recurrence in idiopathic intracranial hypertension: a case-control study. Neurology. 2011 May 3;76(18):1564-7. doi: 10.1212/WNL.0b013e3182190f51. PMID 21536635
- [Background] Aguiar M, Frew E, Mollan SP, Mitchell JL, Ottridge RS, Alimajstorovic Z, Yiangou A, Singhal R, Tahrani AA, Sinclair AJ. The Health Economic Evaluation of Bariatric Surgery Versus a Community Weight Management Intervention Analysis from the Idiopathic Intracranial Hypertension Weight Trial (IIH:WT). Life (Basel). 2021 Apr 30;11(5):409. doi: 10.3390/life11050409. PMID 33946177
- [Background] Elliot L, Frew E, Mollan SP, Mitchell JL, Yiangou A, Alimajstorovic Z, Ottridge RS, Wakerley BR, Thaller M, Grech O, Singhal R, Tahrani AA, Harrison M, Sinclair AJ, Aguiar M. Cost-effectiveness of bariatric surgery versus community weight management to treat obesity-related idiopathic intracranial hypertension: evidence from a single-payer healthcare system. Surg Obes Relat Dis. 2021 Jul;17(7):1310-1316. doi: 10.1016/j.soard.2021.03.020. Epub 2021 Mar 30. PMID 33952427
- [Background] Mahendran V, Ricart P, Levine F, White E, Abolghasemi-Malekabadi K, Williams M, Wadley MS, Perry A, Robinson SJ. Bariatric Surgery as a Viable Treatment for Idiopathic Intracranial Hypertension: a Case Series and Review of Literature. Obes Surg. 2021 Oct;31(10):4386-4391. doi: 10.1007/s11695-021-05587-4. Epub 2021 Jul 28. PMID 34322839
- [Background] Mollan SP, Mitchell JL, Ottridge RS, Aguiar M, Yiangou A, Alimajstorovic Z, Cartwright DM, Grech O, Lavery GG, Westgate CSJ, Vijay V, Scotton W, Wakerley BR, Matthews TD, Ansons A, Hickman SJ, Benzimra J, Rick C, Singhal R, Tahrani AA, Brock K, Frew E, Sinclair AJ. Effectiveness of Bariatric Surgery vs Community Weight Management Intervention for the Treatment of Idiopathic Intracranial Hypertension: A Randomized Clinical Trial. JAMA Neurol. 2021 Jun 1;78(6):678-686. doi: 10.1001/jamaneurol.2021.0659. PMID 33900360
- [Background] Westgate CSJ, Markey K, Mitchell JL, Yiangou A, Singhal R, Stewart P, Tomlinson JW, Lavery GG, Mollan SP, Sinclair AJ. Increased systemic and adipose 11beta-HSD1 activity in idiopathic intracranial hypertension. Eur J Endocrinol. 2022 Jul 4;187(2):323-333. doi: 10.1530/EJE-22-0108. Print 2022 Aug 1. PMID 35584002
- [Background] Abu-Abeid A, Bendayan A, Tome J, Lessing Y, Eldar SM, Keidar A, Dayan D. Long Term Effects of Metabolic and Bariatric Surgery on Idiopathic Intracranial Hypertension. Obes Surg. 2023 Aug;33(8):2615-2619. doi: 10.1007/s11695-023-06696-y. Epub 2023 Jun 23. PMID 37351765
- [Background] Okida LF, Salimi T, Aleman R, Funes DR, Frieder J, Gutierrez D, Montorfano L, Lo Menzo E, Szomstein S, Rosenthal RJ. Midterm benefits of metabolic surgery on symptom remission and medication use in patients with pseudotumor cerebri. Surgery. 2023 Apr;173(4):904-911. doi: 10.1016/j.surg.2022.11.031. Epub 2022 Dec 20. PMID 36549974
- [Background] Kupersmith MJ, Gamell L, Turbin R, Peck V, Spiegel P, Wall M. Effects of weight loss on the course of idiopathic intracranial hypertension in women. Neurology. 1998 Apr;50(4):1094-8. doi: 10.1212/wnl.50.4.1094. PMID 9566400
- [Background] Greener DL, Akarca D, Durnford AJ, Ewbank F, Buckland GR, Hempenstall J. Idiopathic Intracranial Hypertension: Shunt Failure and the Role of Obesity. World Neurosurg. 2020 May;137:e83-e88. doi: 10.1016/j.wneu.2020.01.040. Epub 2020 Jan 16. PMID 31954904
- [Background] Wong R, Madill SA, Pandey P, Riordan-Eva P. Idiopathic intracranial hypertension: the association between weight loss and the requirement for systemic treatment. BMC Ophthalmol. 2007 Sep 21;7:15. doi: 10.1186/1471-2415-7-15. PMID 17888152
- [Background] Sinclair AJ, Burdon MA, Nightingale PG, Ball AK, Good P, Matthews TD, Jacks A, Lawden M, Clarke CE, Stewart PM, Walker EA, Tomlinson JW, Rauz S. Low energy diet and intracranial pressure in women with idiopathic intracranial hypertension: prospective cohort study. BMJ. 2010 Jul 7;341:c2701. doi: 10.1136/bmj.c2701. PMID 20610512
- [Background] Weil R, Kovacs B, Miller N, McDermott MP, Wall M, Kupersmith M, Pi-Sunyer FX; NORDIC Idiopathic Intracranial Hypertension Study Group. A 6-month telephone-based weight loss intervention in overweight and obese subjects with idiopathic intracranial hypertension. Obes Sci Pract. 2016 Apr 5;2(2):95-103. doi: 10.1002/osp4.34. eCollection 2016 Jun. PMID 29071096
- [Background] Koc F, Isik MR, Sefi-Yurdakul N. Weight reduction for a better visual outcome in idiopathic intracranial hypertension. Arq Bras Oftalmol. 2018 Jan-Feb;81(1):18-23. doi: 10.5935/0004-2749.20180006. PMID 29538589
- [Background] Wall M, Johnson CA, Cello KE, Zamba KD, McDermott MP, Keltner JL; NORDIC Idiopathic Intracranial Hypertension Study Group. Visual Field Outcomes for the Idiopathic Intracranial Hypertension Treatment Trial (IIHTT). Invest Ophthalmol Vis Sci. 2016 Mar;57(3):805-12. doi: 10.1167/iovs.15-18626. PMID 26934136
- [Background] Kilgore KP, Lee MS, Leavitt JA, Mokri B, Hodge DO, Frank RD, Chen JJ. Re-evaluating the Incidence of Idiopathic Intracranial Hypertension in an Era of Increasing Obesity. Ophthalmology. 2017 May;124(5):697-700. doi: 10.1016/j.ophtha.2017.01.006. Epub 2017 Feb 7. PMID 28187976
- [Background] Subramaniam S, Fletcher WA. Obesity and Weight Loss in Idiopathic Intracranial Hypertension: A Narrative Review. J Neuroophthalmol. 2017 Jun;37(2):197-205. doi: 10.1097/WNO.0000000000000448. PMID 27636748
- [Background] Tuta S. Cerebral Venous Outflow Implications in Idiopathic Intracranial Hypertension-From Physiopathology to Treatment. Life (Basel). 2022 Jun 8;12(6):854. doi: 10.3390/life12060854. PMID 35743885
- [Background] Raper DMS, Ding D, Buell TJ, Crowley RW, Starke RM, Liu KC. Effect of Body Mass Index on Venous Sinus Pressures in Idiopathic Intracranial Hypertension Patients Before and After Endovascular Stenting. Neurosurgery. 2018 Apr 1;82(4):555-561. doi: 10.1093/neuros/nyx186. PMID 28431144
- [Background] Rajasekharan C, Renjith SW, Marzook A, Parvathy R. Idiopathic intracranial hypertension as the initial presentation of systemic lupus erythematosus. BMJ Case Rep. 2013 Jan 31;2013:bcr2012007886. doi: 10.1136/bcr-2012-007886. PMID 23376664
- [Background] Kilgore KP, Lee MS, Leavitt JA, Frank RD, McClelland CM, Chen JJ. A Population-Based, Case-Control Evaluation of the Association Between Hormonal Contraceptives and Idiopathic Intracranial Hypertension. Am J Ophthalmol. 2019 Jan;197:74-79. doi: 10.1016/j.ajo.2018.09.014. Epub 2018 Sep 21. PMID 30248310
- [Background] Bruce BB, Kedar S, Van Stavern GP, Monaghan D, Acierno MD, Braswell RA, Preechawat P, Corbett JJ, Newman NJ, Biousse V. Idiopathic intracranial hypertension in men. Neurology. 2009 Jan 27;72(4):304-9. doi: 10.1212/01.wnl.0000333254.84120.f5. Epub 2008 Oct 15. PMID 18923135
- [Background] Faz G, Butler IJ, Koenig MK. Incidence of papilledema and obesity in children diagnosed with idiopathic ''benign'' intracranial hypertension: case series and review. J Child Neurol. 2010 Nov;25(11):1389-92. doi: 10.1177/0883073810364853. Epub 2010 Mar 31. PMID 20357237
- [Background] Ardissino M, Moussa O, Tang A, Muttoni E, Ziprin P, Purkayastha S. Idiopathic intracranial hypertension in the British population with obesity. Acta Neurochir (Wien). 2019 Feb;161(2):239-246. doi: 10.1007/s00701-018-3772-9. Epub 2018 Dec 18. PMID 30564882
- [Background] Brara SM, Koebnick C, Porter AH, Langer-Gould A. Pediatric idiopathic intracranial hypertension and extreme childhood obesity. J Pediatr. 2012 Oct;161(4):602-7. doi: 10.1016/j.jpeds.2012.03.047. Epub 2012 May 26. PMID 22633290
- [Background] Paley GL, Sheldon CA, Burrows EK, Chilutti MR, Liu GT, McCormack SE. Overweight and obesity in pediatric secondary pseudotumor cerebri syndrome. Am J Ophthalmol. 2015 Feb;159(2):344-52.e1. doi: 10.1016/j.ajo.2014.11.003. Epub 2014 Nov 7. PMID 25447107
- [Background] Ybarra M, Santos TJD, Queiroz ES, Rachid L, Franco RR, Cominato L, Moura FC, Velhote MC, Damiani D. BARIATRIC SURGERY AS A TREATMENT FOR IDIOPATHIC INTRACRANIAL HYPERTENSION IN A MALE ADOLESCENT: CASE REPORT. Rev Paul Pediatr. 2020 Jan 13;38:e2018239. doi: 10.1590/1984-0462/2020/38/2018239. eCollection 2020. PMID 31939513
- [Background] Zafar S, Panthangi V, Cyril Kurupp AR, Raju A, Luthra G, Shahbaz M, Almatooq H, Foucambert P, Esbrand FD, Khan S. A Systematic Review on Whether an Association Exists Between Adolescent Obesity and Idiopathic Intracranial Hypertension. Cureus. 2022 Aug 16;14(8):e28071. doi: 10.7759/cureus.28071. eCollection 2022 Aug. PMID 36127965
- [Background] Keltner JL, Johnson CA, Cello KE, Wall M; NORDIC Idiopathic Intracranial Hypertension Study Group. Baseline visual field findings in the Idiopathic Intracranial Hypertension Treatment Trial (IIHTT). Invest Ophthalmol Vis Sci. 2014 Apr 29;55(5):3200-7. doi: 10.1167/iovs.14-14243. PMID 24781936
- [Background] Wall M, Hart WM Jr, Burde RM. Visual field defects in idiopathic intracranial hypertension (pseudotumor cerebri). Am J Ophthalmol. 1983 Nov;96(5):654-69. doi: 10.1016/s0002-9394(14)73425-7. PMID 6638133
- [Background] Hoffmann J, Mollan SP, Paemeleire K, Lampl C, Jensen RH, Sinclair AJ. European headache federation guideline on idiopathic intracranial hypertension. J Headache Pain. 2018 Oct 8;19(1):93. doi: 10.1186/s10194-018-0919-2. PMID 30298346
- [Background] Westgate CSJ, Israelsen IME, Jensen RH, Eftekhari S. Understanding the link between obesity and headache- with focus on migraine and idiopathic intracranial hypertension. J Headache Pain. 2021 Oct 10;22(1):123. doi: 10.1186/s10194-021-01337-0. PMID 34629054